CLINICAL TRIAL: NCT03796689
Title: The PCORnet Blood Pressure Home Monitoring Study
Acronym: BP Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-254-53
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Smartphone-linked (Experimental)
  Interventions: Device: Smartphone-linked HBPM and associated app
- Standard (Active Comparator)
  Interventions: Device: Standard HBPM

INTERVENTIONS:
Device: Smartphone-linked HBPM and associated app — Participants in the Smartphone-linked arm of the study will receive an Omron 786N Home Blood Pressure Monitor (HBPM) that can be linked to the Omron Connect app via Bluetooth. They will also receive instructions about how to use their device and download the app and will be provided with publicly available guidelines for HBPM. Participants will be instructed to use their device and app to take readings which they can track over time and share with their provider using the app.
  Arms: Smartphone-linked
Device: Standard HBPM — Participants in the Standard arm of the study will receive an Omron 785N Home Blood Pressure Monitor (HBPM), instructions about how to use their device and publicly available guidelines for HBPM. They will be instructed to use their device to take readings which they can track over time and share with their provider.
  Arms: Standard

SUMMARY:
The PCORnet Blood Pressure Home Monitoring (BP HOME) Study is a patient-level randomized controlled trial that will compare the effectiveness of home blood pressure monitoring (HPBM) with versus without a linked Smartphone application ("app") for helping patients with uncontrolled hypertension achieve a reduction in systolic blood pressure. The trial will be conducted within the National Patient-Centered Clinical Research Network (PCORnet), which supports a research network that enables distributed querying of EHR data in a common data model. It will also use the Eureka Research Platform, an online research platform hosted by UCSF that supports eConsent, online surveys, and data collection from devices such as HBPMs. Data from these two data sources will be used together to accomplish the study aims. Given that HBPM is the guideline-recommended standard of care (without specification of Smartphone linkage), the HPBM devices and the app are all commercially available and currently in use, and that clinicians, with input from patients, will maintain full control of how BP is clinically managed, we believe participation in the project poses minimal risk to participants.

DETAILED DESCRIPTION:
We have designed a patient-level randomized controlled trial that will compare the effectiveness of Smartphone-linked versus standard HBPM for helping patients with uncontrolled hypertension achieve a reduction in their Systolic Blood Pressure (SBP), and patient satisfaction with the device. Our original plan was to recruit 2000 patients who would be randomized in a 1:1 ratio to receive a Smartphone-linked or standard HBPM. However, to recruit higher diversity with more African Americans and LatinX patients, we extended the recruitment period.* We will use data from the electronic health record (EHR), an online patient portal, and the home BP monitor (in the Smartphone-linked arm) to collect outcome data for a period of at least 6 months (for the primary outcome), and up to 18 months (for secondary outcomes, depending on enrollment date). The primary BP control outcome will be reduction in SBP, by clinic measurements, at 6 months. The primary patient satisfaction outcome will be the Net Promoter Score derived from self-reported likelihood of recommending the device to a friend, at 6 months.

*edited after completing recruitment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* At least one ambulatory visit in one of the participating study sites during the past year
* SBP > 145 mmHg at most recent clinic visit (may be treated with BP meds already or not)
* A self-reported commitment to "work on lowering your blood pressure by 10 points or more to reduce your risk of heart attack and stroke"
* Owns a Smartphone (Android or iOS)
* Willing to receive text messages from the study
* Can read/write English well enough to use English-based Smartphone apps and fill out online surveys in English

Exclusion Criteria:

* Has an arm circumference <22 cm or >42 cm
* Owns a functioning HPBM and has used it in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2238 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pletcher, MD MPH, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - University of Florida Health, Gainesville, Florida
  - University Medical Center, New Orleans, Louisiana
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Background] Hamilton DF, Lane JV, Gaston P, Patton JT, Macdonald DJ, Simpson AH, Howie CR. Assessing treatment outcomes using a single question: the net promoter score. Bone Joint J. 2014 May;96-B(5):622-8. doi: 10.1302/0301-620X.96B5.32434. PMID 24788496
- [Background] Krol MW, de Boer D, Delnoij DM, Rademakers JJ. The Net Promoter Score--an asset to patient experience surveys? Health Expect. 2015 Dec;18(6):3099-109. doi: 10.1111/hex.12297. Epub 2014 Oct 27. PMID 25345554
- [Result] Pletcher MJ, Fontil V, Modrow MF, Carton T, Chamberlain AM, Todd J, O'Brien EC, Sheer A, Vittinghoff E, Park S, Orozco J, Lin F, Maeztu C, Wozniak G, Rakotz M, Shay CM, Cooper-DeHoff RM. Effectiveness of Standard vs Enhanced Self-measurement of Blood Pressure Paired With a Connected Smartphone Application: A Randomized Clinical Trial. JAMA Intern Med. 2022 Oct 1;182(10):1025-1034. doi: 10.1001/jamainternmed.2022.3355. PMID 35969408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting screening criteria were invited to participate by mail, email, phone, patient portal message or in person, and directed to the online study portal for eligibility assessment. The first participant was enrolled on August 15, 2019 and the last participant was enrolled on December 31, 2020.
Pre-assignment Details: 137 participants who withdrew consent prior to randomization or did not complete their baseline surveys were excluded.
Period: Overall Study
Arm/Group | Smartphone-linked | Standard
Started | 1051 | 1050
Completed | 1051 | 1050
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smartphone-linked | Standard | Total
Number analyzed (Participants) | 1051 | 1050 | 2101
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13) | 58 (13) | 58 (13)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex, male | 462 | 448 | 910
  Sex, female | 589 | 602 | 1191
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic Asian | 6 | 22 | 28
  Race/Ethnicity: Non-Hispanic Black | 239 | 226 | 465
  Race/Ethnicity: Non-Hispanic White | 676 | 666 | 1342
  Race/Ethnicity: Hispanic/LatinX, any race | 79 | 101 | 180
  Race/Ethnicity: Non-Hispanic, other/multiple races | 51 | 35 | 86
Subjective Social Status [Mean (Standard Deviation); unit: units on a scale] — MacArthur Subjective Social Scale, 1-10 scale (10 = Best off; 1 = Worst off)
  units on a scale | 6.2 (2.2) | 6.2 (2.2) | 6.2 (2.2)
Eligibility systolic BP [Mean (Standard Deviation); unit: mmHg] | 157 (11) | 158 (12) | 157 (11)
Eligibility diastolic BP [Mean (Standard Deviation); unit: mmHg] | 88 (11) | 88 (12) | 88 (12)
Satisfaction with BP management [Mean (Standard Deviation); unit: units on a scale] — 1-5 scale (1 = Very Unsatisfied; 5 = Very Satisfied)
  units on a scale
    Overall | 3.8 (1.1) | 3.7 (1.2) | 3.8 (1.2)
    Your healthcare provider | 4.3 (1.1) | 4.3 (1.0) | 4.3 (1.0)
    Your BP medications | 3.7 (1.2) | 3.7 (1.2) | 3.7 (1.2)
Comfort using technology like a computer or smartphone [Mean (Standard Deviation); unit: units on a scale] — 1-5 scale (1 = Not at all comfortable; 5 = Very comfortable)
  units on a scale | 4.1 (1.1) | 4.1 (1.1) | 4.1 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change is defined by the absolute difference between the SBP measured at the most recent outpatient clinical encounter at the time of enrollment, and the SBP measured at the most recent outpatient clinical encounter 6 months after enrollment. If more than 1 measurement is recorded during a single clinical encounter, the lower/lowest will be used.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Smartphone-linked | Standard
Number analyzed (Participants) | 1051 | 1050
mmHg | 10.8 (18) | 10.6 (18)

2. Primary Outcome: Net Promoter Score
Description: This score is assessed by asking a single question about likelihood of recommending the device to a friend, with options from 1-10 (10 being extremely likely). As per published methods, persons indicating 9 or 10 are considered "Promoters"; persons indicating 7 or 8 are "Passives"; and persons indicating 1-6 are "Detractors". The score is calculated by taking the percent of Promoters and subtracting the percent of Detractors, yielding a score for each group ranging from -100 to 100, with higher scores indicating a better outcome.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smartphone-linked | Standard
Number analyzed (Participants) | 1051 | 1050
score on a scale | 59 (2.81) | 57 (4.00)

ADVERSE EVENTS:
Time Frame: Not applicable: adverse events were not collected.
Description: Adverse events were not collected.
Arm/Group | Smartphone-linked | Standard
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT03796689/Prot_SAP_000.pdf